CLINICAL TRIAL: NCT02581085
Title: Tocotrienol Against the Progression of End Stage Liver Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chandan Sen (Other)
Collaborators: Malaysia Palm Oil Board (Other Government); Indiana University (Other)
Responsible Party: Sponsor-Investigator, Chandan Sen, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1807361301; 136352 (Other: USFDA)
Record Dates: First submitted 2015-06-26; First posted 2015-10-20 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: End Stage Liver Disease; NASH - Nonalcoholic Steatohepatitis; NAFLD - Nonalcoholic Fatty Liver Disease
Keywords: Tocotrienol; Vitamin E
MeSH Terms: conditions — End Stage Liver Disease; Non-alcoholic Fatty Liver Disease | interventions — Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Vehicle (Placebo Comparator): Subjects will take 2 placebo capsules following AM meal, 2 placebo capsules following PM capsules
  Interventions: Other: Placebo
- Tocotrienol supplement (Active Comparator): Subjects will take (2) 200 mg TCT capsules following AM meal, (2) 200 mg TCT following PM meal
  Interventions: Drug: Tocotrienol (TCT)

INTERVENTIONS:
Drug: Tocotrienol (TCT) — TCT is a natural vitamin E supplement with a long history of safe dietary consumption in humans. The objective of the current trial is to validate the outcome observed in an earlier trial that oral TCT attenuates the rise in MELD score over time in patients with end stage liver disease/cirrhosis.
  Arms: Tocotrienol supplement
Other: Placebo — Control study capsule that includes no study product (Vitamin E - Tocotrienol)
  Other Names: vehicle
  Arms: Placebo Vehicle

SUMMARY:
The purpose of this Phase 2 trial is to validate the outcome observed in a previous trial that oral Tocotrienol (TCT) attenuates the rise in MELD score over time in patients with end stage liver disease / cirrhosis. The study is double blind and participants will be randomized to take 2 capsules of TCT (200mg) or placebo twice a day for 3 years.

DETAILED DESCRIPTION:
Tocotrienol (TCT) is a natural vitamin E supplement with a long history of safe dietary consumption. Prior studies with Vitamin E have shown beneficial effects in patients with non-alcoholic fatty liver disease and cirrhosis. The primary purpose of this Phase 2 trial is to validate the outcome observed in an earlier trial that oral TCT attenuates the rise in MELD (Model For End-Stage Liver Disease) score over time in patients with cirrhosis. Outcomes of this trail will direct the design of a future larger multi-center trial.

Study participation will last 3 years. Subjects will be seen for an initial visit, at which consent will be obtained and baseline labs drawn, followed by a Randomization visit 2-14 days later after MELD criteria have been confirmed. If the acceptable labs have not been drawn per standard of care to calculate a MELD score within 90 days before the initial visit, the subject will complete the initial visit as planned, but will then return for a repeat lab draw 60 days later to confirm MELD criteria for eligibility before continuing to the randomization visit.

Enrollment occurs when a subject meets all criteria and is randomized into one of the treatment groups. Subjects will then be seen in the research office by research personnel at 1 week, 2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months, 1 year, 18 months, 2 years, and 3 years. Subject compliance with supplements will be closely followed, as compliance is critical for accurate data. Given the small sample size, subjects who are less than 75% compliant at two consecutive study visits will be discontinued from the study. Subjects will be discontinued if their MELD score increases by more than 25% between 2 consecutive visits or if they receive an organ transplant. Subjects will be declared lost to follow-up (LTFU) if a study visit is unable to be scheduled and completed after 4 documented attempts to contact a subject with no response. In this circumstance, a certified letter will be mailed to the subject's last known address; if no response is received, the subject is LTFU. All subjects discontinued or LTFU before the end of 1 year of study participation will be replaced (see protocol to review study visit activities that will occur). At the Randomization Visit, enrolled subjects will be randomized into one of two treatment groups in a 1:1 manner. Group 1: Placebo vehicle; (2) placebo capsules following AM meal, (2) placebo capsules following PM meal Group 2: 800mg TCT; (2) 200mg TCT capsules following AM meal, (2) 200mg TCT capsules following PM meal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of above, male or female
* ESLD patients with clinically- diagnosed NAFLD or NASH
* Absence of any other possible cause for liver dysfunction
* Stable MELD score of at least 8, but no greater than 17 with <25% change in MELD over the past 60 days prior to enrollment (*Total number of patients with MELD of 8-9 or MELD of 16-17 cannot exceed 40% of cohort)
* Able to speak and understand English
* Willing and able to provide informed consent
* Willing and able to return for regularly scheduled research study visits & comply with study requirements

Exclusion Criteria:

1. Rapid deterioration of liver function, as defined by an increase in MELD score ≥25% over the past 60 days prior to enrollment
2. Hepatocellular carcinoma
3. Positive HIV/AIDS, or other chronic immunodeficiency
4. Concurrent hepatitis B or C infection
5. Current drug and/or alcohol abuse (per treating physician)
6. Bacterial infection at time of enrollment
7. Daily use of dedicated vitamin E supplementation (greater than 100 IU per day) within the 3 months prior to study participation
8. Platelets <35,000 cells/µL, neutrophils <1000 cells/µL, hemoglobin <10g/dL, total bilirubin >3mg/dL, serum creatinine >2.0mg/dL
9. Women who are pregnant, breastfeeding, or plan to become pregnant during course of study participation (36 months)
10. Other significant comorbidities which limit the subject's life expectancy to less than 36 months
11. Concurrent enrollment in another interventional clinical trial
12. ALT >250 U/L
13. AST > 250 U/L
14. Hemoglobin A1C ≥ 9.5 %
15. History of liver transplantation
16. Current or history of HCC
17. Any weight reduction surgery in the preceding 2 years prior to screening or planned surgery during the study
18. Malignancy within 5 years of screening with the exception of a Adequately treated carcinoma in situ of the cervix b. Adequately treated basal or squamous cell cancer or other localized non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of Oral tocotrienols (TCT) on Model for End-Stage Liver Disease (MELD) score. | 3 years
  Lab tests to calculate MELD score will be taken at baseline study visit and the last study visit ( Study visit 17 - 3 years) to see if Oral TCT will significantly attenuate the rise in MELD score over time in patients with End Stage Liver Disease / Cirrhosis

SECONDARY OUTCOMES:
Key Secondary Outcome | 3 yrs
  Composite clinical endpoint defined as any event of all-cause mortality, liver transplant, new onset ascites, hepatic encephalopathy, gastroesophageal variceal hemorrhage, and confirmed increase of MELD score by 3 points due to liver disease.
Change in Child-Pugh Score | 3 years
  change in Child-Pugh Score
Change in ALT Alanine transaminase | 3 years
  Change in ALT (Alanine transaminase)
Events of hepatic decompensation | 3 yrs
  Events of hepatic decompensation
New onset ascites requiring treatment with or without paracentesis | 3 yrs
  New onset ascites requiring treatment with or without paracentesis
GI bleed attributed to variceal bleeding | 3 yrs
  GI bleed attributed to variceal bleeding, requires evaluation by an endoscopy
Hepatic encephalopathy requiring treatment | 3 yrs
  Hepatic encephalopathy requiring treatment, Grade 2 or above according to West Haven Criteria
Need for Liver transplant | 3 yrs
  Need for liver transplant
Death | 3 yrs
  did death occur
Liver fibrosis | 3 yrs
  Liver fibrosis as measured by change in LSM by vibration-controlled transient elastography
Adverse events | 3 yrs
  Did any AEs occur

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, Ph.D, Study Chair — University of Pittsburgh; Raj Vuppalanchi, M.D., Principal Investigator — Indiana Unviersity School of Medicine
Locations (1):
- IU Health Unviersity Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Patel V, Rink C, Gordillo GM, Khanna S, Gnyawali U, Roy S, Shneker B, Ganesh K, Phillips G, More JL, Sarkar A, Kirkpatrick R, Elkhammas EA, Klatte E, Miller M, Firstenberg MS, Chiocca EA, Nesaretnam K, Sen CK. Oral tocotrienols are transported to human tissues and delay the progression of the model for end-stage liver disease score in patients. J Nutr. 2012 Mar;142(3):513-9. doi: 10.3945/jn.111.151902. Epub 2012 Feb 1. PMID 22298568
- [Background] Chitturi S, Abeygunasekera S, Farrell GC, Holmes-Walker J, Hui JM, Fung C, Karim R, Lin R, Samarasinghe D, Liddle C, Weltman M, George J. NASH and insulin resistance: Insulin hypersecretion and specific association with the insulin resistance syndrome. Hepatology. 2002 Feb;35(2):373-9. doi: 10.1053/jhep.2002.30692. PMID 11826411
- [Background] Ray K. NAFLD-the next global epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):621. doi: 10.1038/nrgastro.2013.197. No abstract available. PMID 24185985
- [Background] Schwenger KJ, Allard JP. Clinical approaches to non-alcoholic fatty liver disease. World J Gastroenterol. 2014 Feb 21;20(7):1712-23. doi: 10.3748/wjg.v20.i7.1712. PMID 24587650
- [Background] Schwimmer JB, Behling C, Newbury R, Deutsch R, Nievergelt C, Schork NJ, Lavine JE. Histopathology of pediatric nonalcoholic fatty liver disease. Hepatology. 2005 Sep;42(3):641-9. doi: 10.1002/hep.20842. PMID 16116629
- [Background] Review Team; LaBrecque DR, Abbas Z, Anania F, Ferenci P, Khan AG, Goh KL, Hamid SS, Isakov V, Lizarzabal M, Penaranda MM, Ramos JF, Sarin S, Stimac D, Thomson AB, Umar M, Krabshuis J, LeMair A; World Gastroenterology Organisation. World Gastroenterology Organisation global guidelines: Nonalcoholic fatty liver disease and nonalcoholic steatohepatitis. J Clin Gastroenterol. 2014 Jul;48(6):467-73. doi: 10.1097/MCG.0000000000000116. No abstract available. PMID 24921212
- [Background] Khanna S, Patel V, Rink C, Roy S, Sen CK. Delivery of orally supplemented alpha-tocotrienol to vital organs of rats and tocopherol-transport protein deficient mice. Free Radic Biol Med. 2005 Nov 15;39(10):1310-9. doi: 10.1016/j.freeradbiomed.2005.06.013. PMID 16257640
- [Background] Khanna S, Rink C, Ghoorkhanian R, Gnyawali S, Heigel M, Wijesinghe DS, Chalfant CE, Chan YC, Banerjee J, Huang Y, Roy S, Sen CK. Loss of miR-29b following acute ischemic stroke contributes to neural cell death and infarct size. J Cereb Blood Flow Metab. 2013 Aug;33(8):1197-206. doi: 10.1038/jcbfm.2013.68. Epub 2013 May 1. PMID 23632968
- [Background] Khanna S, Roy S, Slivka A, Craft TK, Chaki S, Rink C, Notestine MA, DeVries AC, Parinandi NL, Sen CK. Neuroprotective properties of the natural vitamin E alpha-tocotrienol. Stroke. 2005 Oct;36(10):2258-64. doi: 10.1161/01.STR.0000181082.70763.22. Epub 2005 Sep 15. PMID 16166580
- [Background] Park HA, Kubicki N, Gnyawali S, Chan YC, Roy S, Khanna S, Sen CK. Natural vitamin E alpha-tocotrienol protects against ischemic stroke by induction of multidrug resistance-associated protein 1. Stroke. 2011 Aug;42(8):2308-14. doi: 10.1161/STROKEAHA.110.608547. Epub 2011 Jun 30. PMID 21719775
- [Background] Patel V, Khanna S, Roy S, Ezziddin O, Sen CK. Natural vitamin E alpha-tocotrienol: retention in vital organs in response to long-term oral supplementation and withdrawal. Free Radic Res. 2006 Jul;40(7):763-71. doi: 10.1080/10715760600672491. PMID 16984003
- [Background] Rink C, Christoforidis G, Khanna S, Peterson L, Patel Y, Khanna S, Abduljalil A, Irfanoglu O, Machiraju R, Bergdall VK, Sen CK. Tocotrienol vitamin E protects against preclinical canine ischemic stroke by inducing arteriogenesis. J Cereb Blood Flow Metab. 2011 Nov;31(11):2218-30. doi: 10.1038/jcbfm.2011.85. Epub 2011 Jun 15. PMID 21673716
- [Background] Gopalan Y, Shuaib IL, Magosso E, Ansari MA, Abu Bakar MR, Wong JW, Khan NA, Liong WC, Sundram K, Ng BH, Karuthan C, Yuen KH. Clinical investigation of the protective effects of palm vitamin E tocotrienols on brain white matter. Stroke. 2014 May;45(5):1422-8. doi: 10.1161/STROKEAHA.113.004449. Epub 2014 Apr 3. PMID 24699052
- [Background] Khosla P, Patel V, Whinter JM, Khanna S, Rakhkovskaya M, Roy S, Sen CK. Postprandial levels of the natural vitamin E tocotrienol in human circulation. Antioxid Redox Signal. 2006 May-Jun;8(5-6):1059-68. doi: 10.1089/ars.2006.8.1059. PMID 16771695
- [Background] Mahipal A, Klapman J, Vignesh S, Yang CS, Neuger A, Chen DT, Malafa MP. Pharmacokinetics and safety of vitamin E delta-tocotrienol after single and multiple doses in healthy subjects with measurement of vitamin E metabolites. Cancer Chemother Pharmacol. 2016 Jul;78(1):157-65. doi: 10.1007/s00280-016-3048-0. Epub 2016 Jun 8. PMID 27278668
- [Background] Mangialasche F, Solomon A, Kareholt I, Hooshmand B, Cecchetti R, Fratiglioni L, Soininen H, Laatikainen T, Mecocci P, Kivipelto M. Serum levels of vitamin E forms and risk of cognitive impairment in a Finnish cohort of older adults. Exp Gerontol. 2013 Dec;48(12):1428-35. doi: 10.1016/j.exger.2013.09.006. Epub 2013 Oct 7. PMID 24113154
- [Background] Meganathan P, Jabir RS, Fuang HG, Bhoo-Pathy N, Choudhury RB, Taib NA, Nesaretnam K, Chik Z. A new formulation of Gamma Delta Tocotrienol has superior bioavailability compared to existing Tocotrienol-Rich Fraction in healthy human subjects. Sci Rep. 2015 Sep 1;5:13550. doi: 10.1038/srep13550. PMID 26323969
- [Background] Springett GM, Husain K, Neuger A, Centeno B, Chen DT, Hutchinson TZ, Lush RM, Sebti S, Malafa MP. A Phase I Safety, Pharmacokinetic, and Pharmacodynamic Presurgical Trial of Vitamin E delta-tocotrienol in Patients with Pancreatic Ductal Neoplasia. EBioMedicine. 2015 Nov 14;2(12):1987-95. doi: 10.1016/j.ebiom.2015.11.025. eCollection 2015 Dec. PMID 26844278